CLINICAL TRIAL: NCT06268821
Title: The Effect on HbA1c of the Initiation of Continuous Glucose Monitoring in Adults With Type 2 Diabetes Treated With Basal Insulin in Finland
Brief Title: Effect on HbA1c of the Initiation of CGM in Adults With Type 2 Diabetes Treated With Basal Insulin in Finland
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Abbott Diabetes Care (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ADC-UK-PMS-23059
Record Dates: First submitted 2024-02-13; First posted 2024-02-20 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Type 2 Diabetes Treated With Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Other): FreeStyle Libre 2 Flash Glucose Monitoring System
  Interventions: Device: FreeStyle Libre 2 Flash Glucose Monitoring System

INTERVENTIONS:
Device: FreeStyle Libre 2 Flash Glucose Monitoring System — Glucose sensors to be worn continuously for 3 months with data used to monitor and manage diabetes treatment and to inform lifestyle choices (diet and exercise)

SUMMARY:
The goal of this clinical study is to determine the impact of starting the use of the FreeStyle Libre 2 glucose monitoring system, over a three month period, on HbA1c in adults with type 2 diabetes treated with a basal insulin regimen.

DETAILED DESCRIPTION:
This is a post-market, multi-centre, prospective, interventional single arm study in Finland.

Participants will use the FreeStyle Libre 2 Flash Glucose Monitoring System, according to the labelling, to monitor their glucose for approximately 3 months. Additional therapies may be introduced, if clinically indicated, based on review of the participant's clinical data and in line with national guidance.

HbA1c will be tested at the start and end of the study for primary endpoint analysis.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 to ≤ 75 years.
* Type 2 diabetes diagnosis ≥1 year prior to enrolment.
* Type 2 diabetes treated with a basal insulin injection regimen with or without other antihyperglycaemic therapy at enrolment.
* Current glucose lowering treatment regimen has been established for at least 3 months prior to enrolment.
* Screening HbA1c ≥59 mmol/mol to ≤108 mmol/mol (≥7.5% and ≤12.0%, inclusive), within the last 60 days.

Exclusion Criteria:

* Participant is currently prescribed prandial or pre-mixed (biphasic) insulin at enrolment.
* Currently participating in another study that could affect glucose measurements or glucose management.
* Currently receiving dialysis treatment or receives dialysis during the study.
* A female participant who is pregnant.
* A breastfeeding female participant.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2024-04-02 (Actual); Primary Completion 2024-07-12 (Actual); Study Completion 2024-07-12 (Actual)

PRIMARY OUTCOMES:
HbA1c | 3 months
  Change in HbA1c within group from baseline

SECONDARY OUTCOMES:
Time in range (TIR) | 3 months
  Time spent in glucose target range (TIR) 3.9 to 10.0 mmol/L (70 to 180 mg/dL)
Time above range (TAR) | 3 months
  Time spent above glucose target range (TAR) >10.0 mmol/L, >13.9 mmol/L and >16.7 mmol/L (>180 mg/dL, >250 mg/dL and >300 mg/dL).
Time below range (TBR) | 3 months
  Time spent below glucose target range (TBR) <3.9 mmol/L and <3.0 mmol/L (<70 mg/dL and <54 mg/dL).
Frequency of hypoglycaemia events | 3 months
  CGM detected hypoglycaemia events defined as ≥15 minutes duration with glucose <3.9mmol/L (<70mg/dL)

CONTACTS AND LOCATIONS:
Overall Officials: Henri Honka, MD, PhD, Principal Investigator — Pihlajalinna, Jämsä
Locations (2):
- Finland (2):
  - Pihlajalinna Jämsä, Välikatu 1,, Jämsä
  - Pihlajalinna Koskiklinikka, Hatanpäänvaltatie 1,, Tampere

IPD SHARING:
Plan to Share IPD: No